CLINICAL TRIAL: NCT02481050
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of Eribulin Mesylate Administered Biweekly (Q2W) for Subjects With Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Metastatic Breast Cancer
Brief Title: Study to Evaluate the Efficacy and Safety of Eribulin Mesylate Administered Biweekly (Q2W) for Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-M001-216
Record Dates: First submitted 2015-06-17; First posted 2015-06-25 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Eribulin Mesylate; Human Epidermal Growth Factor Receptor 2; Metastatic Breast Cancer; HER2-Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Eribulin Mesylate (Experimental): Participants with metastatic HER2-negative breast cancer previously treated with 2 to 5 chemotherapy regimens.
  Interventions: Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin Mesylate will be administered as a 1.4 mg/m2 intravenous (IV) injection over 2 to 5 minutes biweekly on Day 1 and Day 15 of each 28-day cycle.
  Other Names: Halaven, E7389

SUMMARY:
This is a Phase 2, open-label, single arm, multicenter, 2-stage study of eribulin mesylate administered biweekly at 1.4 mg/m2 intravenously for the treatment of participants with HER2-negative metastatic breast cancer previously treated with 2 to 5 chemotherapy regimens.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, single arm, multicenter, 2-stage study of eribulin mesylate administered biweekly at 1.4 mg/m2 intravenously for the treatment of participants with HER2-negative metastatic breast cancer previously treated with 2 to 5 chemotherapy regimens. The study will be conducted in 3 Phases: a Pretreatment Phase (screening visit), a Treatment Phase (starting with Cycle 1 Day 1), and a Posttreatment Phase (End of treatment visit and survival follow up). Participants may remain on study drug as long as they demonstrate clinical benefit or until intercurrent illness, unacceptable toxicity, or disease progression occurs, until the participant withdraws consent, or death.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological adenocarcinoma of the breast.
2. Females, aged greater than or equal to 18 years at time of informed consent.
3. HER2-negative as determined by fluorescence in situ hybridization (FISH); or 0 or 1+ by immunohistochemistry (IHC) staining .
4. Participants with metastatic breast cancer who have received at least 2 and not more than 5 prior chemotherapy regimens.
5. Participants with at least one measurable lesion greater than or equal to 10 mm in the longest diameter for a non-lymph node or greater than or equal to 15 mm in the short-axis diameter for a lymph node as determined by investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
6. Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2.
7. Life expectancy of greater than or equal to 3 months.
8. Any neuropathy must recover to Grade less than or equal to 2 prior to enrollment.
9. Adequate renal function as evidenced by serum creatinine less than or equal to 1.5 mg/dL or calculated creatinine clearance greater than or equal to 50 mL/minute according to the Cockcroft and Gault formula.
10. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than or equal to 1.5 X 10^9/L, hemoglobin greater than or equal to 10.0 g/dL (can be corrected by growth factor or transfusion), and platelet count greater than or equal to 100 X 10^9/L.
11. Adequate liver function as evidenced by total bilirubin less than or equal to 1.5 X upper limit of normal (ULN), alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 X ULN (less than or equal to 5 X ULN in the case of liver metastases), unless there are bone metastases, in which case liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase.
12. Are willing and able to comply with all aspects of the treatment protocol.
13. Provide written informed consent.

Exclusion Criteria:

1. Previous treatment with eribulin.
2. Hypersensitivity to eribulin/excipients or halichondrin B or known intolerance of eribulin.
3. Current enrollment in another clinical study or used of any investigational drug or device within the past 28 days preceding informed consent.
4. Previous treatment with chemotherapy, radiation, biological, or targeted therapy within the last 2 weeks or 5 X half-life, whichever is longer, preceding informed consent.
5. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin ([B-hCG] test). A separate Baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
6. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
7. Females of childbearing potential who had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period or for 28 days after study drug discontinuation.

   Females who are currently abstinent and do not agree to use a double barrier method as described above or to refrain from sexual activity during the study period or for 28 days after study drug discontinuation.

   Females who are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study or for 28 days after study drug discontinuation.
8. Known central nervous system (CNS) disease, except for those participants with treated brain metastasis who are stable for at least 1 month with no evidence of progression or hemorrhage after treatment and no ongoing requirement for corticosteroids.
9. Known human immunodeficiency virus (HIV) positive.
10. Existing anticancer, therapy-related toxicities of Grades greater than or equal to 2, with the exception of alopecia.
11. A prior malignancy other than carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated greater than 5 years previously with no subsequent evidence of recurrence.
12. Clinically significant cardiovascular impairment (congestive heart failure of New York Heart Association [NYHA] Classification greater than II, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia).
13. Clinically significant ECG abnormality, including a marked Baseline prolonged QT/QTc interval (ie, a repeated demonstration of a QTc interval greater than 500 milliseconds).
14. Pulmonary lymphangitic involvement that resulted in pulmonary dysfunction requiring active treatment, including the use of oxygen.
15. History of concomitant medical condition(s) that, in the opinion of the investigator, would compromise the participant's ability to safely complete the study.
16. The investigator's belief that the participant is medically unfit to receive eribulin or unsuitable for any other reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Misir, Study Director — Eisai Inc.
Locations (12):
- United States (12):
  - Facility #1, Denver, Colorado
  - Facility #1, Columbia, Maryland
  - Facility #1, Omaha, Nebraska
  - Facility #1, Albany, New York
  - Facility #1, Portland, Oregon
  - Facility #1, Dallas, Texas
  - Facility #2, Dallas, Texas
  - Facility #1, Houston, Texas
  - Facility #1, San Antonio, Texas
  - Facility #1, Tyler, Texas
  - Facility #1, Leesburg, Virginia
  - Facility #1, Winchester, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in the United States from 16 June 2015 to 05 September 2017.
Pre-assignment Details: A total of 74 participants were screened, of which 16 were screen failures and 58 were randomized to receive study treatment.
Groups:
- Eribulin Mesylate 1.4 mg/m^2: Participants with histologically confirmed human epidermal growth factor receptor 2 (HER2)-negative metastatic breast cancer (MBC) who were previously treated with 2 to 5 chemotherapy regimens received eribulin mesylate 1.4 milligram per square meter (mg/m^2), intravenous infusion over 2 to 5 minutes on Day 1 and Day 15 of each 28-days treatment cycle until intercurrent illness, unacceptable toxicity, disease progression occurred, or until the participant withdrew consent (up to 16 cycles).
Period: Overall Study
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Started | 58
Completed | 0
Not Completed | 58
Not completed — Adverse Event | 1
Not completed — Disease Progression | 47
Not completed — Withdrawal by Subject | 7
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received any amount of study drug.
Groups:
- Eribulin Mesylate 1.4 mg/m^2: Participants with histologically confirmed HER2-negative MBC who were previously treated with 2 to 5 chemotherapy regimens received eribulin mesylate 1.4 mg/m^2, intravenous infusion over 2 to 5 minutes on Day 1 and Day 15 of each 28-days treatment cycle until intercurrent illness, unacceptable toxicity, disease progression occurred, or until the participant withdrew consent (up to 16 cycles).
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 45
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Investigator Assessment
Description: ORR was defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) measured by response evaluation criteria in solid tumors (RECIST) 1.1. CR defined as disappearance of all target lesions (a short diameter is less than [<] 10 millimeter [mm] if it exists in a lymph node). PR defined as at least 30 percent (%) decrease in the sum of the long diameter (LD) of all target lesions, as compared with Baseline summed LD.
Time Frame: From first dose of study drug until intercurrent illness, unacceptable toxicity, disease progression, or until the participant withdrew consent (approximately up to 2.3 years)
Population: The evaluable analysis set (EAS) included all participants who had both an evaluable baseline tumor assessment and an evaluable postbaseline tumor assessment, unless the participants discontinued because of disease progression or toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 57
percentage of participants | 12.3 [5.08 to 23.68]

2. Primary Outcome: Disease Control Rate (DCR) by Investigator Assessment
Description: DCR was defined as the percentage of participants who had BOR of CR, PR, or stable disease (SD) measured by RECIST 1.1. CR defined as disappearance of all target lesions (a short diameter is <10 mm if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the LD of all target lesions, as compared with Baseline summed LD. SD defined as reduction in tumor volume of less than 50% or an increase in the volume of 1 or more measurable lesions of less than 25% without the appearance of any new lesions which was neither tumor shrinkage corresponding to PR nor tumor expansion corresponding to disease progression. SD must be achieved at greater than equal to (>=) 7 weeks after the first eribulin administration to be considered BOR.
Time Frame: as for outcome 1
Population: The EAS included all participants who had both an evaluable baseline tumor assessment and an evaluable postbaseline tumor assessment, unless the participants discontinued because of disease progression or toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 57
percentage of participants | 64.9 [51.13 to 77.09]

3. Secondary Outcome: Progression-Free Survival (PFS) by Investigator Assessment
Description: PFS was defined as the time from date of first dose of study drug to the date of disease progression or death, whichever occurred first.
Time Frame: as for outcome 1
Population: The FAS included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 58
months | 3.6 [2.86 to 4.07]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of first dose of study drug until date of death from any cause.
Time Frame: From date of first dose of study drug administration until date of death from any cause (approximately up to 2.3 years)
Population: The FAS included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 58
months | 12.9 [9.76 to 16.56]

5. Secondary Outcome: Feasibility Rate
Description: Feasibility rate is defined as the percentage of participants completing the first 2 and 4 cycles (1 cycle = 28 days) of eribulin mesylate treatment (4 and 8 doses) without requiring dose delay greater than (>) 5 days or reduction due to adverse event (AE).
Time Frame: Cycle 2 Day 28 and Cycle 4 Day 28 ( cycle length=28 days)
Population: The FAS included all participants who received any amount of study drug. The FAS where data at specified timepoints was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 58
percentage of participants
  First 2 cycles: number analyzed (Participants) | 53
  First 2 cycles | 69.8 [55.7 to 81.7]
  First 4 cycles: number analyzed (Participants) | 22
  First 4 cycles | 50.0 [28.2 to 71.8]

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug (Baseline) up to 30 days after last dose of study drug (approximately up to 2.3 years)
Population: The FAS included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 58
Participants
  TEAE | 58
  SAE | 14

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Baseline) up to 30 days after last dose of study drug (approximately up to 2.3 years)
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
All-Cause Mortality (participants affected / at risk) | 40/58
Serious Adverse Events (participants affected / at risk) | 14/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate 1.4 mg/m^2 (N=58)
Constipation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Pain (General disorders) | 1
Sepsis (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Paraesthesia (Nervous system disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate 1.4 mg/m^2 (N=58)
Anaemia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Eyelids pruritus (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 7
Ocular hyperaemia (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 14
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 6
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Loose tooth (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 17
Stomatitis (Gastrointestinal disorders) | 14
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 2
Chills (General disorders) | 3
Early satiety (General disorders) | 2
Face oedema (General disorders) | 1
Fatigue (General disorders) | 32
Gait disturbance (General disorders) | 3
Localised oedema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 8
Pain (General disorders) | 2
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 7
Cholelithiasis (Hepatobiliary disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 2
Bronchitis viral (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Hordeolum (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Skin bacterial infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 6
Arthropod bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 8
Fibula fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood pressure diastolic decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 22
Platelet count decreased (Investigations) | 2
Troponin increased (Investigations) | 1
Weight decreased (Investigations) | 5
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Amnesia (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 7
Hypoaesthesia (Nervous system disorders) | 4
Neuralgia (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 19
Peroneal nerve palsy (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Device occlusion (Product Issues) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Panic attack (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Bladder prolapse (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 29
Blister (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin tightness (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 3
Thrombosis (Vascular disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lip pain (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes